CLINICAL TRIAL: NCT05776693
Title: Relationships Among Physical and Psychological Status, Social Support, Resource Utilization, Supportive Care Needs in Patients With Gynecological Cancer
Status: Enrolling by invitation | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202210084RINA
Record Dates: First submitted 2022-12-06; First posted 2023-03-20 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Gynecologic Cancer
Keywords: Gynecologic Cancer; Supportive need; Social resource; Social support

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
With the advancement of medical treatments and under the trend of prolonging the survival rate of gynecological cancer patients, the use of social resources and the need for supportive care are particularly important! In the past, studies on patients with gynecological cancer focused on the relation between physical and mental symptoms, intimate relationships, social support, and quality of life. There were few studies on the relationship between social support, resource utilization, and supportive care needs for this group of patients. Therefore, this study research will be conducted on these topics. The results of the study can confirm the current situation of gynecological cancer patients using social resources and the related factors that affect their supportive care needs, and can provide important empirical data for future social resource services and international research design content.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed by a physician as a patient with gynecological cancer
* Aged 20 or above, with clear consciousness and able to communicate in Mandarin and Taiwanese.
* After reading the consent form, accept the questionnaire.

Exclusion Criteria:

* Unconscious and unable to communicate verbally to complete the interview for this study

Ages: 20 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Because the research object is gynecological cancer patient, it must be a person with a female physiological structure.
Study Population: Patients who have diagnosed gynecological cancer.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-11-24 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Supportive Care Needs Survey. | 1 time points: From date of approaching patient until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months.
  Patients' supportive care needs by Supportive Care Needs Survey.It is a 5-Point Likert Scale,higher scores mean more care needs.

SECONDARY OUTCOMES:
Physical and Psychological Symptoms Scale | 1 time points: From date of approaching patient until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months.
  Patients' physical and psychological symptoms will be measured by Physical and Psychological Symptom Scale.It use Numerical Rating Scale(VRS)0-10.It is a 11 Point Likert Scale(e. g. 0 is no pain; 10 is unbearable pain) .
Medical Outcomes Study Social Support Survey. | 1 time points: From date of approaching patient until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months.
  Patients' social support by Medical Outcomes Study Social Support Survey(MOS-SSS).It is a 5 Point Likert Scale(0-5) ,higher scores represents receiving more social support.
Social resource assessment . | 1 time points: From date of approaching patient until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months.
  Patients' utilization of social resource assessment scale developed by the research team. It is a 5 Point Likert Scale(0-5).The higher the score, the more frequently the resource is used.Also answer how helpful and useful the resource is(0-10),higher scores represents more helpful and useful.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University, Taipei, Taiwan